CLINICAL TRIAL: NCT03888976
Title: Cholecystoduodenal Fistula With and Without Gallstone Ileus: A Case Series
Brief Title: Cholecystoduodenal Fistula With and Without Gallstone Ileus
Status: Completed | Type: Observational
Sponsor: Tecnologico de Monterrey (Other)
Responsible Party: Sponsor
Other Study IDs: CDF031
Record Dates: First submitted 2019-03-20; First posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Gallbladder Diseases
Keywords: Cholecystoduodenal fistula; Gallbladder
MeSH Terms: conditions — Gallbladder Diseases; Intestinal Fistula | interventions — Cholecystectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cholecystectomy — Cholecystectomy with repair of duodenal wall.

SUMMARY:
Observative and descriptive study of 10 patients, which were diagnosed with a Cholecystoduodenal fistula, All electronic medical records were retrospectively reviewed.

DETAILED DESCRIPTION:
A cholecystoenteric fistula is an uncommon complication of gallstone disease, although most studies in the English literature concern biliary-enteric fistulas. The aim of this study was to present a case series of patients with a cholecystoduodenal fistula (CDF), with or without gallstone ileus, along with the surgical outcomes.

From 2015 to 2018, 3245 consecutive patients underwent cholecystectomy for gallbladder disease at our institution, of whom 10 were diagnosed with a CDF. All electronic medical records were retrospectively reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cholecystoduodenal fistula

Exclusion Criteria:

* Patients with cholecystocolonic fistula or cholecystogastric fistula

Ages: 15 Years to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent surgical resection of cholecystoduodenal fistula
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-03-03 (Actual)

PRIMARY OUTCOMES:
Median Age | Feb 01- 2020
  Age in years
Median value of white blood count | Feb 01-2020
  It will presented in cells/L
Type of surgery performed | Feb 01-2020
  It will described the type of procedure, either conventional or laparoscopic
Surgical complications | Feb 01-2020
  Morbidity will be described as Yes or No
Recovering time | Feb 01-2020
  The median time in days, after the procedure and full recovery of the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Metropolitano, San Nicolás de los Garza, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No
not apply